CLINICAL TRIAL: NCT00484900
Title: Open Randomized Multi-Centre Trial, Comparing Artesunate-Sulfamethoxypyrazine-Pyrimethamine FDC Over 3 Days, Artesunate-Sulfamethoxypyrazine-Pyrimethamine FDC Over 48 Hours and Artemether-Lumefantrine FDC Over 3 Days on P. Falciparum Malaria
Brief Title: Multi-Centre Trial Comparing Three Artemisinin-Based Combination Treatments on P. Falciparum Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dafra Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005/57/01
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2007-06

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Open randomized multi-centre clinical trial in Africa; Uncomplicated P. falciparum malaria; Artemisinin-based Combination Therapy; Artesunate + sulfalene + pyrimethamine; 24 hour treatment; Artemether + lumefantrine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Co-Arinate FDC
Drug: Coartem

SUMMARY:
The purpose of this open randomised multi-centre clinical trial is to test the hypothesis that three pills of the fixed dose combination artesunate/sulfamethoxypyrazine/pyrimethamine, administered over 24 hours is not inferior in efficacy to the same drug administered over 48 hours and that the fixed dose combination artesunate/sulfamethoxypyrazine/pyrimethamine As/SMP fdc, independently of the duration of its dose interval, is not inferior in efficacy to 6 - 24 pills (number of pills administered to respectively children and adults)of the 60 hours treatment of artemether/lumefantrine for the treatment of uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* age at least 6 months,
* weight at least 5 kg,
* residing in one of the four countries (Mali, Cameroon, Sudan, Rwanda),
* able to receive oral treatment,
* having an axillary body temperature of more than 37,5 degrees Celsius or history of fever within the proceeding 24 hours,
* suffering from a mono specific P. falciparum infection with a parasite density between 2000 and 200000 asexual forms per micro litre of blood.

Exclusion Criteria:

* presence of severe or complicated malaria (WHO 2000),
* severe concomitant pathology or one that needs a medical follow-up incompatible with the study,
* allergic to one of the drugs involved in this study,
* pregnant (reported pregnancy, detected clinically or with the β HCG test),
* use of one of the anti-malaria drugs involved in this study during 28 days preceding inclusion.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1390 (Actual)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
PCR corrected Adequate Clinical and Parasitological Response | on day 28 (follow-up period)
Early treatment failure | between day 0 and day 3
Late clinical failure | between day 4 and day 28
Late parasitological failure | between day 7 and day 28

SECONDARY OUTCOMES:
Parasitic clearance | 28 day follow-up period
Fever clearance | 28 day follow-up period
Parasitological re-infection | 28 day follow-up period
Gametocyte carriage | 28 day follow-up period
Safety - Adverse events | 28 day follow-up period
Haemoglobin levels | 28 day follow-up period
Clinical and biological tolerance (Haemogram + Lever tests) | 28 day follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Issaka Sagara, Dr, Principal Investigator — University of Bamako, Mali; Wilfred F Mbacham, Dr, Principal Investigator — University Yaoundé, Cameroon; Ishag A Adam, Dr, Principal Investigator — University of Khartoum, Sudan; Stephen Rulisa, Dr, Principal Investigator — Kigali Central University Hospital, Rwanda
Locations (4):
- Cameroon Baptist Convention Clinic of Biyem-Assi, Yaoundé, Cameroon
- Health centres of Samako, Kolle and Bancoumane, Bamako, Mali
- Health centres Rwamagana and Muhima, Kigali, Rwanda
- Alhara Alola Health centre, New Halfa, Sudan

REFERENCES:
- [Derived] Sagara I, Rulisa S, Mbacham W, Adam I, Sissoko K, Maiga H, Traore OB, Dara N, Dicko YT, Dicko A, Djimde A, Jansen FH, Doumbo OK. Efficacy and safety of a fixed dose artesunate-sulphamethoxypyrazine-pyrimethamine compared to artemether-lumefantrine for the treatment of uncomplicated falciparum malaria across Africa: a randomized multi-centre trial. Malar J. 2009 Apr 14;8:63. doi: 10.1186/1475-2875-8-63. PMID 19366448